CLINICAL TRIAL: NCT00114504
Title: Detection of Atherosclerotic Plaque Inflammation and Visualization of Anti-inflammatory Effects of Statins on Plaque Inflammation by FDG-PET
Brief Title: Detection of Plaque Inflammation by Positron Emission Tomography (PET)-Effects of Simvastatin on Plaque Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Hisashi Kai, Associate professor, Kurume University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KurumeU-2416
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; inflammation; statins; PET; carotid ultrasonography
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin group (Experimental): Patients with FDG-positive plaque who received simvastatin and diet therapy
  Interventions: Drug: simvastatin
- Control group (No Intervention): Patients FDG-positive plaque who received diet therapy alone

INTERVENTIONS:
Drug: simvastatin — simvastatin 5-10 mg/day
  Other Names: control
  Arms: Simvastatin group

SUMMARY:
The purpose of this study is to determine whether FDG-PET is capable of detecting atherosclerotic plaque inflammation and monitoring the effects of statins on plaque inflammation. The usefulness of FDG-PET in risk stratification is also investigated.

DETAILED DESCRIPTION:
There is increasing evidence that inflammation plays a role in progression and destabilization of atherosclerotic plaque. However, currently, no non-invasive method is available for detecting plaque inflammation in clinical practice. FDG-PET can visualize activated metabolic levels of not only tumor cells but also inflammatory cells. Thus, it is possible that FDG-PET can detect atherosclerotic plaque inflammation and that, if so, FDG-PET can monitor the direct effect of statins on plaque inflammation. Additionally, monitoring the plaque inflammation by FDG-PET may be useful for determining the risk stratification of atherosclerotic patients.

Originally, we sought to compare patients with FDG-positive plaque with patients with plaque but not with FDG uptake, patients with FDG-positive plaque receiving statin therapy, and patients with FDG-positive plaque receiving diet management therapy. However, because patient number enrolled in the study was too small, the comparison was performed between FDG-positive patients with and without any statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Protocol 1: patients who had carotid atherosclerosis detected by carotid ultrasound.
* Protocol 2: patients who underwent FDG-PET for cancer screening and had vascular FDG uptakes

Exclusion Criteria:

* Active inflammatory diseases
* Dyslipidemia under medications
* Uncontrolled diabetes mellitus, vasculitis, symptomatic coronary artery disease, symptomatic cerebrovascular diseases
* Known systemic disorders such as hepatic, renal, hematopoietic, and malignant diseases

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09; Primary Completion 2007-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hisashi Kai, MD, PhD, Principal Investigator — The Third Department of Internal Medicine, Kurume University
Locations (1):
- Kurume University Hospital, Kurume, Japan

REFERENCES:
- [Derived] Tahara N, Kai H, Yamagishi S, Mizoguchi M, Nakaura H, Ishibashi M, Kaida H, Baba K, Hayabuchi N, Imaizumi T. Vascular inflammation evaluated by [18F]-fluorodeoxyglucose positron emission tomography is associated with the metabolic syndrome. J Am Coll Cardiol. 2007 Apr 10;49(14):1533-9. doi: 10.1016/j.jacc.2006.11.046. Epub 2007 Mar 26. PMID 17418291

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin Group: Patients with FDG-positive carotid artery and/or aorta who received simvastatin and diet therapy
- Control Group: Patients with FDG-positive carotid artery and/or aorta who received diet therapy alone
Period: Overall Study
Arm/Group | Simvastatin Group | Control Group
Started | 21 | 22
Completed | 21 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin Group | Control Group | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9) | 62 (6) | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 21 | 22 | 43
  No Japanese | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Plaque Inflammation
Description: Change in plaque inflammation was assessed by changes in the plaque SUV.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- Simvastatin Group: Patients with FDG-positive carotid artery and/or aorta who received simvastatin and diet therapy for 3 months
- Control Group: Patients with FDG-positive carotid artery and/or aorta who received diet therapy alone or 3 months
Arm/Group | Simvastatin Group | Control Group
Number analyzed (Participants) | 21 | 22
SUV | 1.59 (0.22) | 1.63 (0.12)

2. Secondary Outcome: Circulating Inflammation Marker
Description: Change in circulating hsCRP levels
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Simvastatin Group Baseline: Patients with FDG-positive carotid artery and/or aorta who received simvastatin and diet therapy at baseline
- Simvastatin Group at 3 Month: Patients with FDG-positive carotid artery and/or aorta who received simvastatin and diet therapy for 3 months
- Control Group Baseline: Patients with FDG-positive carotid artery and/or aorta who received diet therapy alone at baseline
- Control Group at 3 Months: Patients with FDG-positive carotid artery and/or aorta who received diet therapy alone for 3 months.
Arm/Group | Simvastatin Group Baseline | Simvastatin Group at 3 Month | Control Group Baseline | Control Group at 3 Months
Number analyzed (Participants) | 21 | 21 | 22 | 22
mg/dL | 0.09 (0.11) | 0.06 (0.07) | 0.11 (0.16) | 0.07 (0.06)

ADVERSE EVENTS:
Arm/Group | Simvastatin Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes